CLINICAL TRIAL: NCT02395679
Title: A Phase I Study on Dendritic Cells Loaded With Allogeneous Cell Lysate in Patients With Mesothelioma as Maintenance Treatment After Chemotherapy
Brief Title: Dendritic Cells Loaded With Allogeneous Cell Lysate in Mesothelioma Patients
Acronym: MesoCancerVa
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, joost hegmans, Head production, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL44330.000.14
Record Dates: First submitted 2015-01-30; First posted 2015-03-23 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Mesothelioma
Keywords: Dendritic cell-based immunotherapy
MeSH Terms: conditions — Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MesoCancerVac (Experimental): Autologous dendritic cells loaded with a mixture of 5 allogenic mesothelioma tumor cell lysates 3 to 5 vaccinations with 10x10e6, 25x10e6 or 50x10e6 loaded dendritic cells i.d. and i.v. administration every two weeks
  Interventions: Biological: MesoCancerVac

INTERVENTIONS:
Biological: MesoCancerVac — A leukapheresis is performed of which the monocytes are used for differentiation to DCs using specific cytokines. Pulsed autologous DCs (MesoCancerVac) are re-injected 3 times every two weeks. After the third injection with MesoCancerVac, revaccinations to boost the immune system are given after 3 and 6 months.

SUMMARY:
Malignant mesothelioma is an aggressive pleural disease, related to asbestos exposure. At present, cytotoxic chemotherapy is the only evidence based treatment for the disease, but efficacy is limited. The investigators have shown both in a murine model, as for the first time in patients, that dendritic cell-based immunotherapy induces tumor specific T-cell responses. However the quality and quantity of the autologous tumor cell lysate to load the dendritic cells was a major impediment for these trials. The investigators have now developed a clinical grade allogeneic tumor cell lysate which can be used to load dendritic cells of patients.

DETAILED DESCRIPTION:
Objective: To investigate the safety of an allogeneic tumor cell lysate (PheraLys) loaded onto autologous dendritic cells (MesoCancerVac) in patients with malignant mesothelioma (MM).

Study design: A phase I study with a classical 3*3 design. Study population: Adult patients with malignant mesothelioma who were treated with chemotherapy as standard treatment.

Intervention: After chemotherapy, a leukapheresis is performed of which the monocytes are used for differentiation to DCs using specific cytokines. Pulsed autologous DCs (MesoCancerVac) are re-injected 3 times every two weeks. After the third injection with MesoCancerVac, revaccinations to boost the immune system are given after 3 and 6 months.

Main study parameters/endpoints: The aim of this phase I protocol is to study the toxicity and safety of MesoCancerVac (DC-based immunotherapy) in MM patients. Toxicities will be scored according to common toxicity criteria version 4.0. The following toxicities occurring during 8 weeks after the first vaccination, will be considered as dose-limiting toxicities (DLTs).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients have to undergo extra outdoor visits for this study (10-20) and extra invasive procedures especially for this trial, like a catheter in a blood vessel. These are invasive procedure but risks are limited. This iv entrance is necessary every time, for the leukopheresis, for blood samples and for the injection of the dendritic cells. A leucopheresis is a standard procedure and will be performed according to guidelines. There is a limited risk for transient thrombocytopenia and leukopenia.

The administration of autologous cells, that have been loaded with allogeneic human materials, is a potential risk and that is the subject of the study. Because not the lysate itself is administered to the patients but only when it is processed by the dendritic cells of the patient the investigators expect these risks to be limited.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Patients with histological or cytological confirmed diagnosed ,malignant mesothelioma, who are non progressive after at least 4 cycles of cisplatin and pemetrexed containing chemotherapy (as determined by CT scanning).
* Measurable disease on CT scanning in two dimensions by a radiologic imaging study.
* Patients must be at least 18 years old and must be able to give written informed consent.
* Patients must be ambulatory (WHO performance status 0,1, or 2 [Appendix E&F]) The expected survival must be at least 3 months.
* Patients must have normal organ function and adequate bone marrow reserve: absolute neutrophil count > 1.0 x 10e9/l, platelet count > 100 x 10e9/l, and Hb > 6.0 mmol/l.(as determined during screening
* Positive delayed type hypersensitivity skin test (induration > 2mm after 48 hrs) against at least one positive control antigen tetanus toxoid.
* Ability to return to the Erasmus Medical Center for adequate follow-up as required by this protocol.
* Written informed consent according to good clinical practice
* Planned start date of vaccination between 5 weeks after the last dosage of chemotherapy

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Medical or psychological impediment to probable compliance with the protocol.
* Current use of steroids (or other immunosuppressive agents). Patients must have had 6 weeks of discontinuation and must stop of any such treatment during the time of the study. Prophylactic usage of dexamethasone during chemotherapy is excluded from that 6 weeks interval
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the patient has been disease-free for five years.
* Serious concomitant disease, or active infections.
* History of autoimmune disease or organ allografts, or with active acute or chronic infection, including HIV and viral hepatitis.
* Serious intercurrent chronic or acute illness such as pulmonary (asthma or COPD) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for investigational DC treatment.
* Known allergy to shell fish (may contain KLH).
* Pregnant or lactating women.
* Inadequate peripheral vein access to perform leukapheresis
* Concomitant participation in another clinical trial
* An organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent, and preclude participation in the full protocol and follow-up.
* Absence of assurance of compliance with the protocol. Lack of availability for follow-up assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to establish a tolerable dose of MesoCancerVac in patients with malignant mesothelioma | 4 weeks after third administration
  Tolerability of MesoCancerVac is monitored by performing clinical laboratory tests (autoimmune responses), assessments of vital signs, full clinical examination, occurrence of adverse events.

SECONDARY OUTCOMES:
The secondary objective is the evaluation of an immune response after MesoCancerVac | 2 months after third administration
  Immune response is evaluated by measuring :
  The functionality of T-cells by laboratory testing (cytotoxicity and interferon-gamma secretion)

CONTACTS AND LOCATIONS:
Overall Officials: Henk C Hoogsteden, MD PhD, Study Director — Erasmus Medical Center Cancer Institure
Locations (1):
- Erasmus MC, Dept. of Pulmonary Medicine, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Background] Hegmans JP, Veltman JD, Lambers ME, de Vries IJ, Figdor CG, Hendriks RW, Hoogsteden HC, Lambrecht BN, Aerts JG. Consolidative dendritic cell-based immunotherapy elicits cytotoxicity against malignant mesothelioma. Am J Respir Crit Care Med. 2010 Jun 15;181(12):1383-90. doi: 10.1164/rccm.200909-1465OC. Epub 2010 Feb 18. PMID 20167848
- [Result] Cornelissen R, Heuvers ME, Maat AP, Hendriks RW, Hoogsteden HC, Aerts JG, Hegmans JP. New roads open up for implementing immunotherapy in mesothelioma. Clin Dev Immunol. 2012;2012:927240. doi: 10.1155/2012/927240. Epub 2012 Jun 24. PMID 22778767
- [Result] Cornelissen R, Lievense LA, Heuvers ME, Maat AP, Hendriks RW, Hoogsteden HC, Hegmans JP, Aerts JG. Dendritic cell-based immunotherapy in mesothelioma. Immunotherapy. 2012 Oct;4(10):1011-22. doi: 10.2217/imt.12.108. PMID 23148753
- [Result] Hegmans JP, Hemmes A, Aerts JG, Hoogsteden HC, Lambrecht BN. Immunotherapy of murine malignant mesothelioma using tumor lysate-pulsed dendritic cells. Am J Respir Crit Care Med. 2005 May 15;171(10):1168-77. doi: 10.1164/rccm.200501-057OC. Epub 2005 Mar 11. PMID 15764728
- [Derived] van Gulijk M, Belderbos B, Dumoulin D, Cornelissen R, Bezemer K, Klaase L, Dammeijer F, Aerts J. Combination of PD-1/PD-L1 checkpoint inhibition and dendritic cell therapy in mice models and in patients with mesothelioma. Int J Cancer. 2023 Apr 1;152(7):1438-1443. doi: 10.1002/ijc.34293. Epub 2022 Oct 3. PMID 36104949
- [Derived] Vroman H, Balzaretti G, Belderbos RA, Klarenbeek PL, van Nimwegen M, Bezemer K, Cornelissen R, Niewold ITG, van Schaik BD, van Kampen AH, Aerts JGJV, de Vries N, Hendriks RW. T cell receptor repertoire characteristics both before and following immunotherapy correlate with clinical response in mesothelioma. J Immunother Cancer. 2020 Mar;8(1):e000251. doi: 10.1136/jitc-2019-000251. PMID 32234848